CLINICAL TRIAL: NCT02521285
Title: Effect of Aspirin on Biomarkers of Barrett's Esophagus After Successful Eradication of Barrett's Esophagus With Radiofrequency Ablation
Brief Title: Aspirin in Preventing Disease Recurrence in Patients With Barrett Esophagus After Successful Elimination by Radiofrequency Ablation
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NCI-2015-01265; NCI-2015-01265 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2013-0819; N01-CN-2012-00034; HHSN261201200034I; 2015-0819 (Other: M D Anderson Cancer Center); MDA2013-02-02 (Other: DCP); N01CN00034 (NIH); P30CA016672 (NIH)
Record Dates: First submitted 2015-08-11; First posted 2015-08-13 (Estimated); Results first posted 2023-05-01 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-09

CONDITIONS: Barrett Esophagus; Esophageal Adenocarcinoma
MeSH Terms: conditions — Barrett Esophagus; Adenocarcinoma Of Esophagus | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (aspirin) (Experimental): Patients receive aspirin PO QD for 12 months.
  Interventions: Drug: Aspirin; Other: Laboratory Biomarker Analysis; Other: Questionnaire Administration
- Arm B (placebo) (Placebo Comparator): Patients receive placebo PO QD for 12 months.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Placebo Administration; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Aspirin — Given PO
  Other Names: Acetylsalicylic Acid; ASA; Aspergum; Ecotrin; Empirin; Entericin; Extren; Measurin
  Arms: Arm A (aspirin)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Placebo Administration — Given PO
  Arms: Arm B (placebo)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized phase II trial studies the safety of and how well aspirin works in preventing Barrett's esophagus from returning after it has been successfully eliminated by radiofrequency ablation. Studying samples of tissue from patients with Barrett's esophagus for the levels of a specific protein that is linked to developing Barrett's esophagus may help doctors learn whether aspirin can prevent it from returning after it has been successfully treated.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To conduct a randomized, double blind, placebo-controlled phase II chemoprevention trial, investigating whether supplementation with aspirin 325 mg/day for 12 months is safe and reduces the expression of CDX2 messenger ribonucleic acid (mRNA) (a biomarker which has been associated with the risk of developing Barrett's esophagus [BE]) in comparison to placebo after successful radiofrequency ablation (RFA).

SECONDARY OBJECTIVES:

I. To assess safety at 12 months. II. To assess differences in the expression of CDX2 at 18 months, activation status of NF-kB by assessing levels of total and phosphorylated (phospho)-p65 and cytoplasmic to nuclear translocation of phospho-p65 which is likely to be affected by aspirin.

III. To assess the prostanoid marker, prostaglandin E2, and prostaglandin synthases, which are known to respond to aspirin and to correlation with clinicopathological factors in the esophageal cancer.

IV. To assess differences in the expression of proinflammatory cytokines known to induce activation of NFkB, i.e., TNFalpha, IL-1beta, IL-6, IL-10, IL-17A, IL-23 will be measured.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM A: Patients receive aspirin orally (PO) once daily (QD) for 12 months.

ARM B: Patients receive placebo PO QD for 12 months.

After completion of study treatment, patients are followed up at 1, 3, 6, 9, 12, and 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Known diagnosis of histologically-confirmed BE with or without dysplasia (as defined by the presence of specialized columnar epithelium anywhere in the tubular esophagus with >= 1 cm of circumferential involvement or non-circumferential involvement of specialized columnar epithelium) requiring radiofrequency ablation
* Documentation of complete ablation of BE after radiofrequency ablation on two endoscopic examinations at least 3 months apart (including no evidence of BE on surveillance biopsies) as determined by the pathologist at each site; completion of ablation should have occurred no greater than 36 months prior to randomization
* The effects of the candidate chemoprevention agents on the developing human fetus remain incompletely defined; for this reason, persons of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a participant become pregnant or suspect she is pregnant while participating in this trial, she should inform the research personnel and her clinical care provider immediately
* Willingness to provide tissue samples for research purposes
* No chronic use of aspirin or nonsteroidal anti-inflammatory drugs (NSAIDs) or selective cyclooxygenase-2 (COX-2) inhibitors during one month prior to randomization; chronic use is defined as any aspirin or NSAID use on >= 7 days during one month preceding the beginning of randomization
* Hemoglobin >= 10 g/dL or hematocrit >= 30% (obtained =< 45 days prior to randomization)
* Leukocyte count >= 3,000/microliter (obtained =< 45 days prior to randomization)
* Platelet count >= 100,000/microliter (obtained =< 45 days prior to randomization)
* Absolute neutrophil count >= 1,500/microliter (obtained =< 45 days prior to randomization)
* Creatinine =< 2.5 x institutional upper limit of normal (ULN) (obtained =< 45 days prior to randomization)
* OR glomerular filtration rate (GFR) > 30 ml/min/1.73 m^2 (obtained =< 45 days prior to randomization)
* Total bilirubin =< 2 x institutional ULN (obtained =< 45 days prior to randomization)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) =< 2.5 x institutional ULN (obtained =< 45 days prior to randomization)
* Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN (obtained =< 45 days prior to randomization)
* A negative serum pregnancy test at baseline, but within 21 days of randomization, for persons of childbearing potential only
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Ability to understand and the willingness to sign a written informed consent document; a legally authorized representative (LAR) may sign informed consent for persons who do not have the capacity to legally consent to take part in the study

Exclusion Criteria:

* Inability to abstain from, NSAID (including aspirin), and selective COX-2 inhibitor therapy at the time of randomization through the completion of the study (the study period is defined as baseline to exit endoscopy at 18 months after randomization which defines the completion of the study); participants may take Tylenol and non-NSAID pain relievers
* Current or planned use of anticoagulant drugs such as: warfarin, heparin, low molecular weight heparin, Plavix, or Aggrenox throughout the course of the study
* Individuals taking the drugs listed below may not be randomized unless they are willing to stop the medications (and possibly change to alternative non-excluded medications to treat the same conditions) no less than 1 month prior to starting aspirin or placebo on this study; consultation with the participant's primary care provider will be obtained prior to stopping any agent; the use of the following drugs or drug classes is prohibited during aspirin/placebo treatment:

  * NSAIDs: such as aspirin, Naprosyn, ketorolac and others NSAIDs
  * COX-2 inhibitors: such as celecoxib, rofecoxib
  * Valproic acid
  * Sulfinpyrazone
  * Probenecid
  * Corticosteroids (other than short-term use defined as less than 2 weeks or pro re nata [prn (when necessary)] use of an inhaler less than twice per month)
  * Platelet aggregation inhibitors, except in a monitored antithrombotic regimen
  * Methotrexate (MTX)
  * Vaccines containing live viruses
  * Gingko
* Individuals with uncontrolled renal insufficiency or renal failure
* Participants with fundoplication within the past year, bariatric surgery or any other major upper gastrointestinal (GI) surgery; fundoplication more than one year ago will not be grounds for exclusion; cholecystectomy will not be grounds for exclusion
* History of invasive cancer diagnosis =< 12 months prior to randomization, excepting nonmelanoma skin cancer; patients with T1a adenocarcinoma of the esophagus arising in the setting of Barrett's esophagus are eligible for enrollment in the trial
* History of cancer treatment =< 12 months prior to randomization, excepting hormonal therapy (except treatment for non-melanoma skin cancer or carcinoma-in-situ of the cervix)
* Receipt of any other investigational agents =< 3 months prior to randomization, except innocuous agents with no known interaction with the study agents (e.g., standard dose multivitamins or topical agents for limited skin conditions), at the discretion of the protocol lead investigator at each participating site
* History of allergic reactions attributed to aspirin or compounds of similar chemical or biologic composition to the study agent
* History of endoscopically or radiographically diagnosed peptic ulcer disease with upper GI bleeding during the past 5 years or history of endoscopically or radiographically diagnosed peptic ulcer disease with upper GI bleeding any time while taking aspirin
* Uncontrolled intercurrent illness including, but not limited to: ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, bleeding disorder, vitamin K deficiency, alcohol abuse (defined as ingestion of 3 or more drinks per day) or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women
* Breast feeding women
* Surveillance biopsies demonstrating residual BE at qualifying exam
* Presence of an esophageal stricture defined as "any recognizable change in esophageal luminal caliber that is accompanied by symptoms of dysphagia, or any asymptomatic narrowing that either will not allow any adult endoscope to pass or allows passage with resistance"
* Patients with human immunodeficiency virus (HIV) infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-01-15 (Actual); Primary Completion 2019-06-18 (Actual); Study Completion 2026-03-17 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Bresalier, Principal Investigator — M.D. Anderson Cancer Center
Locations (10):
- United States (9):
  - UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Northwestern University, Chicago, Illinois
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - M D Anderson Cancer Center, Houston, Texas
- Saint Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Bresalier RS. Chemoprevention of Barrett's Esophagus and Esophageal Adenocarcinoma. Dig Dis Sci. 2018 Aug;63(8):2155-2162. doi: 10.1007/s10620-018-5149-6. PMID 29948566

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 21 participants were randomized due to 12 were unevaluable.
Groups:
- Arm A (Aspirin): Participants received aspirin 325 mg orally (PO) once daily for 12 months
- Arm B (Placebo): Participants received placebo daily
Period: Overall Study
Arm/Group | Arm A (Aspirin) | Arm B (Placebo)
Started | 10 | 11
Completed | 8 | 8
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Aspirin) | Arm B (Placebo) | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 3 | 8
  >=65 years | 5 | 8 | 13
Age, Continuous [Median (Full Range); unit: years] | 64.5 [49 to 78] | 67 [49 to 84] | 67 [49 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 7 | 8 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 11 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 10 | 11 | 21
Baseline cdx2/normalized to GAPDH [Median (Full Range); unit: percentage of biomarker levels] | 0.34 [0.005 to 0.908] | 0.438 [0.064 to 4.537] | 0.384 [0.005 to 4.537]
Baseline p-p65/total p65 corrected for tubulin [Median (Full Range); unit: percentage of biomarker levels] | 0.484 [0.046 to 0.838] | 0.624 [0.108 to 1.916] | 0.484 [0.046 to 1.916]

OUTCOME MEASURES:

1. Primary Outcome: Difference in the Change of CDX2 mRNA Levels in Esophageal Mucosa Between Participants Taking Aspirin and Placebo at 12 Months (Location A)
Description: Measured the absolute and relative values in percentage of biomarker levels CDX2 mRNA levels in the esophageal mucosa at baseline and 12 months for each participant taking aspirin versus placebo at Location A (1 cm above GE Junction.) The difference in the change were measured by the total RNAs were isolated from squamous and neosquamous mucosal biopsy specimens using Trizol and quantitated by spectrophotometry.
Time Frame: Baseline and 12 months
Population: 1 participant withdrew consent and decided to take a baby aspirin, per PCP recommendation in the Aspirin arm and 1 participant was lost to follow up, 1 participant withdrew consent, and 1 participant adverse event in the Placebo arm
Measure: Median (Full Range); unit: change of percentage of CDX2 mRNA levels
Arm/Group | Arm A (Aspirin) | Arm B (Placebo)
Number analyzed (Participants) | 7 | 5
change of percentage of CDX2 mRNA levels
  12 month (Absolute) | 0.01 [-0.82 to 0.82] | -0.1 [-0.57 to 0]
  12 month (Relative) | 0.05 [-0.94 to 2.34] | -0.87 [-0.99 to -0.23]
Statistical Analysis 1: Comparison: Arm A (Aspirin) vs Arm B (Placebo); Test type: Superiority; p = 0.343, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm A (Aspirin) vs Arm B (Placebo); Test type: Superiority; p = 0.149, t-test, 2 sided

2. Primary Outcome: Differences in the Change of CDX2 Messenger Ribonucleic Acid (mRNA) Levels in Esophageal Squamous Tissue Between Participants Taking Aspirin Supplementation Versus Those Taking Placebo (Location B)
Description: Measured the absolute and relative values change in the biomarker levels CDX2 mRNA levels in the esophageal mucosa at baseline and 12 months for each participant taking aspirin versus placebo at Location B (middle of former Barrett's segment). The difference in the change were measured by the total RNAs were isolated from squamous and neosquamous mucosal biopsy specimens using Trizol and quantitated by spectrophotometry.
Time Frame: Baseline and 12 months
Measure: Median (Full Range); unit: change of percentage of CDX2 mRNA levels
Arm/Group | Arm A (Aspirin) | Arm B (Placebo)
Number analyzed (Participants) | 8 | 8
change of percentage of CDX2 mRNA levels
  12 month change (Absolute) | -0.18 [-0.60 to 0] | -0.17 [-4.43 to 0.62]
  12 month change (Relative) | -0.7 [-0.90 to -0.25] | -0.6 [-1.0 to 9.76]
Statistical Analysis 1: Comparison: Arm A (Aspirin) vs Arm B (Placebo); Test type: Superiority; p = 0.878, t-test, 2 sided

3. Primary Outcome: Differences in the Change of CDX2 Messenger Ribonucleic Acid (mRNA) Levels in Esophageal Squamous Tissue Between Participants Taking Aspirin Supplementation Versus Those Taking Placebo ( Location C)
Description: Measured the absolute and relative values change in the biomarker levels CDX2 mRNA levels in the esophageal mucosa at baseline and 12 months for each participant taking aspirin versus placebo at Location C (2 cm above former Barrett's segment). The difference in the change were measured by the total RNAs were isolated from squamous and neosquamous mucosal biopsy specimens using Trizol and quantitated by spectrophotometry.
Time Frame: Baseline and 12 months
Measure: Median (Full Range); unit: change of percentage of CDX2 mRNA levels
Arm/Group | Arm A (Aspirin) | Arm B (Placebo)
Number analyzed (Participants) | 8 | 8
change of percentage of CDX2 mRNA levels
  12 month change (Absolute) | -0.25 [-1.04 to 0.04] | -0.17 [-0.82 to 0.52]
  12 month change (Relative) | -0.98 [-1.00 to 0.95] | -0.51 [-0.90 to 1.45]
Statistical Analysis 1: Comparison: Arm A (Aspirin) vs Arm B (Placebo); Test type: Superiority; p = 0.382, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm A (Aspirin) vs Arm B (Placebo); Test type: Superiority; p = 0.05, t-test, 2 sided

4. Primary Outcome: Differences in the Activation Status of NF-kB by Assessing Levels of Total and Phospho-p65 and Cytoplasmic to Nuclear Translocation of Phospho-p65 at 12 Months (Location A)
Description: Measured the absolute and relative values change in the biomarker levels p-p65/total p65 in the esophageal mucosa at baseline and 12 months for each participant taking aspirin versus placebo at Location A, 1 cm above GE Junction. The difference in the change were measured by using esophageal squamous and neosquamous mucosal biopsies taken before and after treatment with aspirin, levels of phospho-p65 and total p65 were determined by Western blot and quantitated by densitometry.
Time Frame: Baseline and 12 months
Population: as for outcome 1
Measure: Median (Full Range); unit: change of % of p-p65/total p65 levels
Arm/Group | Arm A (Aspirin) | Arm B (Placebo)
Number analyzed (Participants) | 7 | 5
change of % of p-p65/total p65 levels
  12 month change (Absolute) | 0.16 [-0.43 to 1.38] | 0.16 [-1.89 to 0.37]
  12 month change (Relative) | 0.26 [-0.65 to 13.17] | 0.84 [-0.80 to 32.08]
Statistical Analysis 1: Comparison: Arm A (Aspirin) vs Arm B (Placebo); Test type: Superiority; p = 0.53, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm A (Aspirin) vs Arm B (Placebo); Test type: Superiority; p = 1, t-test, 2 sided

5. Primary Outcome: Differences in the Activation Status of NF-kB by Assessing Levels of Total and Phospho-p65 and Cytoplasmic to Nuclear Translocation of Phospho-p65 at 12 Months (Location B)
Description: Measured the absolute and relative values change in the biomarker levels p-p65/total p65 in the esophageal mucosa at baseline and 12 months for each participant taking aspirin versus placebo at Location B (middle of former Barrett's segment)The difference in the change were measured by using esophageal squamous and neosquamous mucosal biopsies taken before and after treatment with aspirin, levels of phospho-p65 and total p65 were determined by Western blot and quantitated by densitometry.
Time Frame: Baseline and 12 months
Measure: Median (Full Range); unit: change of % of p-p65/total p65 levels
Arm/Group | Arm A (Aspirin) | Arm B (Placebo)
Number analyzed (Participants) | 8 | 8
change of % of p-p65/total p65 levels
  12 month change (Absolute) | -0.12 [-0.40 to 1.26] | -0.32 [-1.15 to 0.30]
  12month change (Relative) | -0.37 [-0.82 to 13.37] | -0.57 [-0.95 to 2.80]
Statistical Analysis 1: Comparison: Arm A (Aspirin) vs Arm B (Placebo); Test type: Superiority; p = 0.234, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm A (Aspirin) vs Arm B (Placebo); Test type: Superiority; p = 0.442, t-test, 2 sided

6. Primary Outcome: Differences in the Activation Status of NF-kB by Assessing Levels of Total and Phospho-p65 and Cytoplasmic to Nuclear Translocation of Phospho-p65 at 12 Months (Location C)
Description: Measured the absolute and relative values change in the biomarker levels p-p65/total p65 in the esophageal mucosa at baseline and 12 months for each participant taking aspirin versus placebo at Location C (2 cm above former Barrett's segment). The difference in the change were measured by using esophageal squamous and neosquamous mucosal biopsies taken before and after treatment with aspirin, levels of phospho-p65 and total p65 were determined by Western blot and quantitated by densitometry.
Time Frame: Baseline and 12 months
Measure: Median (Full Range); unit: change of % of p-p65/total p65 levels
Arm/Group | Arm A (Aspirin) | Arm B (Placebo)
Number analyzed (Participants) | 8 | 8
change of % of p-p65/total p65 levels
  12 month change (Absolute) | -0.37 [-0.76 to 0.15] | -0.28 [-0.83 to 0.23]
  12month change (Relative) | -0.53 [-0.77 to 2.56] | -0.6 [-0.88 to 0.20]
Statistical Analysis 1: Comparison: Arm A (Aspirin) vs Arm B (Placebo); Test type: Superiority; p = 0.645, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm A (Aspirin) vs Arm B (Placebo); Test type: Superiority; p = 0.878, t-test, 2 sided

7. Secondary Outcome: Number of Participants With Adverse Events (AE)
Description: Number of Participants experiencing adverse events by maximum grade (grades 1-3). Safety assessed by comparison of adverse events using the NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. AEs will be assessed according to the CTCAE grade associated with the AE term. All adverse events are listed in the Adverse Events Overview.
Time Frame: Up to 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Aspirin) | Arm B (Placebo)
Number analyzed (Participants) | 8 | 8
Participants
  Adverse Event Grade 1 | 5 | 5
  Adverse Event Grade 2 | 2 | 5
  Adverse Event Grade 3 | 5 | 3

8. Secondary Outcome: Differences in the Change of CDX2 mRNA Levels in Esophageal Squamous Tissue Between Participants Taking Aspirin Supplementation Versus Those Taking Placebo at 18 Months (Location A)
Description: Measured the change in the biomarker levels CDX2 mRNA levels in esophageal mucosa at baseline and 18 months for each participant taking aspirin versus placebo at Location A, 1 cm above GE Junction. The difference in the change were measured by the total RNAs will be isolated from squamous and neosquamous mucosal biopsy specimens using Trizol and quantitated by spectrophotometry.
Time Frame: Baseline to 18 months
Measure: Median (Full Range); unit: percentage of biomarkers level
Arm/Group | Arm A (Aspirin) | Arm B (Placebo)
Number analyzed (Participants) | 3 | 1
percentage of biomarkers level | -56 [-86 to 122] | 58 [-86 to 122]

9. Secondary Outcome: Differences in the Change of CDX2 mRNA Levels in Esophageal Squamous Tissue Between Participants Taking Aspirin Supplementation Versus Those Taking Placebo at 18 Months (Location B)
Description: Measured change in the biomarker levels CDX2 mRNA levels in esophageal mucosa at baseline and 18 months for each participant taking aspirin versus placebo at Location B (middle of former Barrett's segment). The difference in the change were measured by the total RNAs will be isolated from squamous and neosquamous mucosal biopsy specimens using Trizol and quantitated by spectrophotometry.
Time Frame: Up to 18 months
Measure: Median (Full Range); unit: percentage of biomarkers level
Arm/Group | Arm A (Aspirin) | Arm B (Placebo)
Number analyzed (Participants) | 4 | 1
percentage of biomarkers level | -45 [-99 to 1218] | -74 [-99 to 1218]

10. Secondary Outcome: Differences in the Change of CDX2 mRNA Levels in Esophageal Squamous Tissue Between Participants Taking Aspirin Supplementation Versus Those Taking Placebo at 18 Months (Location C)
Description: Measured the change in the biomarker levels CDX2 mRNA levels in esophageal mucosa at baseline and 18 months for each participant taking aspirin versus placebo at Location C (2 cm above former Barrett's segment). The difference in the change were measured by the total RNAs will be isolated from squamous and neosquamous mucosal biopsy specimens using Trizol and quantitated by spectrophotometry.
Time Frame: Baseline to 18 months
Measure: Median (Full Range); unit: percentage of biomarkers level
Arm/Group | Arm A (Aspirin) | Arm B (Placebo)
Number analyzed (Participants) | 4 | 1
percentage of biomarkers level | -93 [-99 to -43] | -53 [-99 to -43]

11. Secondary Outcome: Differences in the Activation Status of NF-kB by Assessing Levels of Total and Phospho-p65 and Cytoplasmic to Nuclear Translocation of Phospho-p65 at 18 Months (Location A)
Description: Measured the change in the biomarker levels p-p65/total p65 in the esophageal mucosa at baseline and 18 months for each participant taking aspirin versus placebo at Location A, 1 cm above GE Junction. The difference in the change were measured by using esophageal squamous and neosquamous mucosal biopsies taken before and after treatment with aspirin, levels of phospho-p65 and total p65 were determined by Western blot and quantitated by densitometry.
Time Frame: Baseline up to 18 months
Population: Participants with biopsies available at 18-months.
Measure: Median (Full Range); unit: percentage of biomarkers level
Arm/Group | Arm A (Aspirin) | Arm B (Placebo)
Number analyzed (Participants) | 3 | 1
percentage of biomarkers level | -71 [-94 to 1] | .113 [-94 to 1]

12. Secondary Outcome: Differences in the Activation Status of NF-kB by Assessing Levels of Total and Phospho-p65 and Cytoplasmic to Nuclear Translocation of Phospho-p65 at 18 Months (Location B)
Description: Measured the change in the biomarker levels of p-p65/total p65 in the esophageal mucosa at baseline and 18 months for each participant taking aspirin versus placebo at Location B (middle of former Barrett's segment). The difference in the change were measured by using esophageal squamous and neosquamous mucosal biopsies taken before and after treatment with aspirin, levels of phospho-p65 and total p65 were determined by Western blot and quantitated by densitometry.
Time Frame: Baseline up to 18 months
Measure: Median (Full Range); unit: percentage of biomarkers level
Arm/Group | Arm A (Aspirin) | Arm B (Placebo)
Number analyzed (Participants) | 4 | 1
percentage of biomarkers level | -59 [-91 to 1643] | 393 [-91 to 1643]

13. Secondary Outcome: Differences in the Activation Status of NF-kB by Assessing Levels of Total and Phospho-p65 and Cytoplasmic to Nuclear Translocation of Phospho-p65 at 18 Months (Location C)
Description: Measured the change in the biomarker levels p-p65/total p65 in esophageal mucosa at baseline and 18 months for each participant taking aspirin versus placebo at Location C (2 cm above former Barrett's segment). The difference in the change were measured by using esophageal squamous and neosquamous mucosal biopsies taken before and after treatment with aspirin, levels of phospho-p65 and total p65 were determined by Western blot and quantitated by densitometry.
Time Frame: Baseline up to 18 months
Measure: Median (Full Range); unit: percentage of biomarkers level
Arm/Group | Arm A (Aspirin) | Arm B (Placebo)
Number analyzed (Participants) | 4 | 1
percentage of biomarkers level | -29 [-64 to 16] | .37 [-64 to 16]

14. Secondary Outcome: Differences in the Change of txb2 at 12 Months (Location A)
Description: Measured the absolute and relative values change in the biomarker levels txb2 levels in the esophageal mucosa at baseline and 12 months for each participant taking aspirin versus placebo at Location A, 1 cm above GE Junction. The difference in the change were measured by the Liquid chromatography-mass spectrometry (LC/MS/MS) analyses.
Time Frame: Baseline and 12 months
Measure: Median (Full Range); unit: change of percentage of txb2 levels
Arm/Group | Arm A (Aspirin) | Arm B (Placebo)
Number analyzed (Participants) | 7 | 5
change of percentage of txb2 levels
  12 month change (Absolute) | -2.07 [-8.48 to 2.33] | -1.07 [-51.57 to 3.27]
  12 month change (Relative) | -0.61 [-0.94 to 1.98] | -0.73 [-099 to 206]
Statistical Analysis 1: Comparison: Arm A (Aspirin) vs Arm B (Placebo); Test type: Superiority; p = 0.755, t-test, 2 sided

15. Secondary Outcome: Differences in the Change of tbx2 at 12 Months (Location B)
Description: Measured the absolute and relative values change in the biomarker levels txb2 levels in the esophageal mucosa at baseline and 12 months for each participant taking aspirin versus placebo at Location B (middle of former Barrett's segment). The difference in the change were measured by the Liquid chromatography-mass spectrometry (LC/MS/MS) analyses.
Time Frame: Baseline and 12 months
Measure: Median (Full Range); unit: change of percentage of tbx2 levels
Arm/Group | Arm A (Aspirin) | Arm B (Placebo)
Number analyzed (Participants) | 7 | 8
change of percentage of tbx2 levels
  12 month change (Absolute) | -2.33 [-52.34 to 0.81] | -0.19 [-46.98 to 2.52]
  12 month change (Relative) | -0.69 [-1.00 to .70] | 0.76 [-1.00 to 4.81]
Statistical Analysis 1: Comparison: Arm A (Aspirin) vs Arm B (Placebo); Difference between arms; Test type: Superiority; p = 0.397, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm A (Aspirin) vs Arm B (Placebo); Difference in arms; Test type: Superiority; p = 0.983, t-test, 2 sided

16. Secondary Outcome: Differences in the Change of tbx2 at 12 Months (Location C)
Description: Measured the absolute and relative values change in the biomarker levels txb2 levels in the esophageal mucosa at baseline and 12 months for each participant taking aspirin versus placebo at Location C (2 cm above former Barrett's segment). The difference in the change were measured by the Liquid chromatography-mass spectrometry (LC/MS/MS) analyses.
Time Frame: Baseline and 12 months
Measure: Median (Full Range); unit: change of percentage of tbx2 levels
Arm/Group | Arm A (Aspirin) | Arm B (Placebo)
Number analyzed (Participants) | 8 | 8
change of percentage of tbx2 levels
  12 month change (Absolute) | -3.58 [-16.26 to 1.05] | 0.5 [-30.48 to 5.55]
  12 month change (Relative) | -0.81 [-1.00 to 1.09] | 1.18 [-1.00 to 3.94]
Statistical Analysis 1: Comparison: Arm A (Aspirin) vs Arm B (Placebo); Test type: Superiority; p = 0.065, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm A (Aspirin) vs Arm B (Placebo); Test type: Superiority; p = 0.203, t-test, 2 sided

17. Secondary Outcome: Differences in the Change of pge1 at 12 Months ( Location A)
Description: Measured the absolute and relative values change in the biomarker levels pge1 levels in the esophageal mucosa at baseline and 12 months for each participant taking aspirin versus placebo at A (1 cm above GE Junction). The difference in the change were measured by the Liquid chromatography-mass spectrometry (LC/MS/MS) analyses.
Time Frame: Baseline and 12 months
Measure: Median (Full Range); unit: change of percentage of pge1 levels
Arm/Group | Arm A (Aspirin) | Arm B (Placebo)
Number analyzed (Participants) | 7 | 5
change of percentage of pge1 levels
  12 month change (Absolute) | -2.29 [-16.39 to 2.52] | -1.13 [-44.74 to 2.95]
  12 month change (Relative) | -0.52 [-0.98 to 2.21] | -0.87 [-1.00 to 1.10]
Statistical Analysis 1: Comparison: Arm A (Aspirin) vs Arm B (Placebo); Test type: Superiority; p = 0.755, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm A (Aspirin) vs Arm B (Placebo); Test type: Superiority; p = 0.343, t-test, 2 sided

18. Secondary Outcome: Differences in the Change of pge1 at 12 Months (Location B)
Description: Measured the absolute and relative values change in the biomarker levels pge1 levels in the esophageal mucosa at baseline and 12 months for each participant taking aspirin versus placebo at Location B (middle of former Barrett's segment). The difference in the change were measured by the Liquid chromatography-mass spectrometry (LC/MS/MS) analyses.
Time Frame: Baseline and 12 months
Measure: Median (Full Range); unit: change of percentage of pge1 levels
Arm/Group | Arm A (Aspirin) | Arm B (Placebo)
Number analyzed (Participants) | 7 | 8
change of percentage of pge1 levels
  12 month change (Absolute) | -7.22 [-13.63 to 1.12] | -0.08 [-17.61 to 1.65]
  12 month change (Relative) | -0.73 [-0.95 to 0.72] | -0.19 [-0.97 to 0.62]
Statistical Analysis 1: Comparison: Arm A (Aspirin) vs Arm B (Placebo); Test type: Superiority; p = 0.281, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm A (Aspirin) vs Arm B (Placebo); Test type: Superiority; p = 0.189, t-test, 2 sided

19. Secondary Outcome: Differences in the Change of pge1 at 12 Months (Location C)
Description: Measured the absolute and relative values change in the biomarker levels pge1 levels in the esophageal mucosa at baseline and 12 months for each participant taking aspirin versus placebo at Location C (2 cm above former Barrett's segment). The difference in the change were measured by the Liquid chromatography-mass spectrometry (LC/MS/MS) analyses.
Time Frame: Baseline and 12 months
Measure: Median (Full Range); unit: change of percentage of pge1 levels
Arm/Group | Arm A (Aspirin) | Arm B (Placebo)
Number analyzed (Participants) | 8 | 8
change of percentage of pge1 levels
  12 month change (Absolute) | -7.79 [-40.65 to 7.99] | 2.71 [-19.72 to 18.54]
  12 month change (Relative) | -0.75 [-0.90 to 13.43] | 2.48 [-0.95 to 11.59]
Statistical Analysis 1: Comparison: Arm A (Aspirin) vs Arm B (Placebo); Test type: Superiority; p = 0.083, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm A (Aspirin) vs Arm B (Placebo); Test type: Superiority; p = 0.195, t-test, 2 sided

20. Secondary Outcome: Differences in the Change of pge2 at 12 Months (Location A)
Description: Measured the absolute and relative values change in the biomarker levels pge2 levels in the esophageal mucosa at baseline and 12 months for each participant taking aspirin versus placebo at A (1 cm above GE Junction). The difference in the change were measured by the Liquid chromatography-mass spectrometry (LC/MS/MS) analyses.
Time Frame: Baseline and 12 months
Measure: Median (Full Range); unit: change of percentage of pge2 levels
Arm/Group | Arm A (Aspirin) | Arm B (Placebo)
Number analyzed (Participants) | 7 | 5
change of percentage of pge2 levels
  12 month change (Absolute) | -6.77 [-38.18 to 8.53] | -5.13 [-110.54 to 6.57]
  12 month change (Relative) | -0.24 [-0.96 to 1.83] | -0.78 [-0.92 to 0.58]
Statistical Analysis 1: Comparison: Arm A (Aspirin) vs Arm B (Placebo); Test type: Superiority; p = 0.755, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm A (Aspirin) vs Arm B (Placebo); Test type: Superiority; p = 0.432, t-test, 2 sided

21. Secondary Outcome: Differences in the Change of pge2 at 12 Months (Location B)
Description: Measured the absolute and relative values change in the biomarker levels pge2 levels in the esophageal mucosa at baseline and 12 months for each participant taking aspirin versus placebo at Location B (middle of former Barrett's segment). The difference in the change were measured by the Liquid chromatography-mass spectrometry (LC/MS/MS) analyses.
Time Frame: Baseline and 12 months
Measure: Median (Full Range); unit: change of percentage of pge2 levels
Arm/Group | Arm A (Aspirin) | Arm B (Placebo)
Number analyzed (Participants) | 7 | 8
change of percentage of pge2 levels
  12 month change (Absolute) | -20.53 [-71.98 to 2.46] | -11 [-59.68 to 8.71]
  12 month change (Relative) | -0.74 [-0.95 to 0.27] | -0.51 [-0.95 to 1.08]
Statistical Analysis 1: Comparison: Arm A (Aspirin) vs Arm B (Placebo); Test type: Superiority; p = 0.463, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm A (Aspirin) vs Arm B (Placebo); Test type: Superiority; p = 0.189, t-test, 2 sided

22. Secondary Outcome: Differences in the Change in pge2 at 12 Months (Location C)
Description: Measured the absolute and relative values change in the biomarker levels pge2 levels in the esophageal mucosa at baseline and 12 months for each participant taking aspirin versus placebo at Location C (2 cm above former Barrett's segment). The difference in the change were measured by the Liquid chromatography-mass spectrometry (LC/MS/MS) analyses.
Time Frame: Baseline and 12 months
Measure: Median (Full Range); unit: change of percentage of pge2 levels
Arm/Group | Arm A (Aspirin) | Arm B (Placebo)
Number analyzed (Participants) | 8 | 8
change of percentage of pge2 levels
  12 month change (Absolute) | -19.23 [-85.32 to 19.03] | 9.94 [-155.89 to 43.35]
  12 month change (Relative) | -0.7 [-0.95 to 5.27] | 1.96 [-0.98 to 10.28]
Statistical Analysis 1: Comparison: Arm A (Aspirin) vs Arm B (Placebo); Test type: Superiority; p = 0.105, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm A (Aspirin) vs Arm B (Placebo); Test type: Superiority; p = 0.161, t-test, 2 sided

23. Secondary Outcome: Differences in the Change of a13pge1 at 12 Months (Location A)
Description: Measured the absolute and relative values change in the biomarker levels a13pge1 levels in the esophageal mucosa at baseline and 12 months for each participant taking aspirin versus placebo at Location A (1 cm above GE Junction). The difference in the change were measured by the Liquid chromatography-mass spectrometry (LC/MS/MS) analyses.
Time Frame: Baseline and 12 months
Measure: Median (Full Range); unit: change of percentage of a13pge1 levels
Arm/Group | Arm A (Aspirin) | Arm B (Placebo)
Number analyzed (Participants) | 7 | 5
change of percentage of a13pge1 levels
  Absolute Value | -0.29 [-7.05 to 0.93] | 0 [-5.78 to 4.38]
  Relative Value | -99 [-100 to -83] | -93 [-100 to -86]

24. Secondary Outcome: Differences in the Change of a13pge1 at 12 Months ( Location B)
Description: Measured the absolute and relative values change in the biomarker levels a13pge1 levels in the esophageal mucosa at baseline and 12 months for each participant taking aspirin versus placebo at Location B (middle of former Barrett's segment). The difference in the change were measured by the Liquid chromatography-mass spectrometry (LC/MS/MS) analyses.
Time Frame: Baseline and 12 months
Measure: Median (Full Range); unit: change of percentage of a13pge1 levels
Arm/Group | Arm A (Aspirin) | Arm B (Placebo)
Number analyzed (Participants) | 7 | 8
change of percentage of a13pge1 levels
  12 month change (Absolute) | -1.62 [-10.32 to 0.00] | 0.19 [-6.51 to 0.72]
  12 month change (Relative) | -92 [-100 to -74] | -65 [-65 to -65]

25. Secondary Outcome: Differences in the Change in a13pge1 at 12 Months (Location C)
Description: Measured the absolute and relative values change in the biomarker levels a13pge1 levels in the esophageal mucosa at baseline and 12 months for each participant taking aspirin versus placebo at Location C (2 cm above former Barrett's segment). The difference in the change were measured by the Liquid chromatography-mass spectrometry (LC/MS/MS) analyses.
Time Frame: Baseline and 12 months
Measure: Median (Full Range); unit: change of percentage of a13pge1 levels
Arm/Group | Arm A (Aspirin) | Arm B (Placebo)
Number analyzed (Participants) | 8 | 8
change of percentage of a13pge1 levels
  12 month change (Absolute) | 0 [-3.4 to 0.75] | 0 [-3.83 to 1.01]
  12 month change (Relative | -61 [-100 to 200] | -100 [-100 to -100]
Statistical Analysis 1: Comparison: Arm A (Aspirin) vs Arm B (Placebo); Test type: Superiority; p = 0.518, t-test, 2 sided

26. Secondary Outcome: Differences in the Change of a13pge2 at 12 Months (Location A)
Description: Measured the absolute and relative values change in the biomarker levels a13pge2 levels in the esophageal mucosa at baseline and 12 months for each participant taking aspirin versus placebo at Location A (1 cm above GE Junction). The difference in the change were measured by the Liquid chromatography-mass spectrometry (LC/MS/MS) analyses.
Time Frame: Baseline and 12 months
Measure: Median (Full Range); unit: change of percentage of a13pge2 levels
Arm/Group | Arm A (Aspirin) | Arm B (Placebo)
Number analyzed (Participants) | 7 | 5
change of percentage of a13pge2 levels
  12 month change (Absolute) | -4.25 [-19.76 to 1.79] | -2.23 [-215.45 to 22.72]
  12 month change (Relative) | -0.93 [-1.00 to 1.05] | -0.8 [-1.00 to 7.43]
Statistical Analysis 1: Comparison: Arm A (Aspirin) vs Arm B (Placebo); Test type: Superiority; p = 0.876, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm A (Aspirin) vs Arm B (Placebo); Test type: Superiority; p = 0.505, t-test, 2 sided

27. Secondary Outcome: Differences in the Change of a13pge2 at 12month (Location B)
Description: Measured the absolute and relative values change in the biomarker levels a13pge2 levels in the esophageal mucosa at baseline and 12 months for each participant taking aspirin versus placebo at Location B (middle of former Barrett's segment). The difference in the change were measured by the Liquid chromatography-mass spectrometry (LC/MS/MS) analyses.
Time Frame: Baseline and 12 months
Measure: Median (Full Range); unit: change of percentage of a13pge2 levels
Arm/Group | Arm A (Aspirin) | Arm B (Placebo)
Number analyzed (Participants) | 7 | 8
change of percentage of a13pge2 levels
  12 month change (Absolute) | -13.94 [-85.07 to 0.82] | -5.56 [-169.75 to 2.80]
  12 month change (Relative) | -0.89 [-0.98 to 0.86] | -0.73 [-0.99 to 1.05]
Statistical Analysis 1: Comparison: Arm A (Aspirin) vs Arm B (Placebo); Test type: Superiority; p = 0.463, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm A (Aspirin) vs Arm B (Placebo); Test type: Superiority; p = 0.094, t-test, 2 sided

28. Secondary Outcome: Differences in the Change of a13pge2 at 12 Months (Location C)
Description: Measured the absolute and relative values change in the biomarker levels a13pge2 levels in the esophageal mucosa at baseline and 12 months for each participant taking aspirin versus placebo at Location C (2 cm above former Barrett's segment). The difference in the change were measured by the Liquid chromatography-mass spectrometry (LC/MS/MS) analyses.
Time Frame: Baseline and 12 months
Measure: Median (Full Range); unit: percentage of a13pge2 biomarkers level
Arm/Group | Arm A (Aspirin) | Arm B (Placebo)
Number analyzed (Participants) | 8 | 8
percentage of a13pge2 biomarkers level
  12 month change (Absolute) | -8.18 [-31.56 to 2.42] | 2.78 [-87.29 to 25.17]
  12 month change (Relative) | -0.51 [-1.00 to 5.57] | 2.27 [-0.98 to 11.22]
Statistical Analysis 1: Comparison: Arm A (Aspirin) vs Arm B (Placebo); Test type: Superiority; p = 0.105, t-test, 2 sided
Statistical Analysis 2: Comparison: Arm A (Aspirin) vs Arm B (Placebo); Test type: Superiority; p = 0.13, t-test, 2 sided

29. Other Pre Specified Outcome: Differences in the Prostanoid Marker, Prostaglandin E2, and Prostaglandin Synthases
Description: Listed separately as #7-13 Secondary Outcome Measures.
Time Frame: Baseline up to 18 months
Reporting Status: Not Posted

30. Other Pre Specified Outcome: Differences in the Expression of Proinflammatory Cytokines Known to Induce Activation of NFkB
Time Frame: Baseline up to 18 months
Population: Differences in the Expression of Proinflammatory Cytokines (a secondary endpoint) was not measured as there was insufficient biopsy material to perform these measurements. Alternatively we measured multiple additional prostaglandins and downstream markers as secondary endpoints since we were able to use smaller amounts of sample on a platform which allowed multiple measurements. These results are detailed in section which lists prostanoid measurements.
Arm/Group | Arm A (Aspirin) | Arm B (Placebo)
Number analyzed (Participants) | 0 | 0

31. Other Pre Specified Outcome: Incidence of Barrett's Esophagus (BE) Recurrence
Time Frame: Baseline up to 18 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: baseline and at each visit throughout the trial (including Month 1, every 3 months by phone calls and/or mail interviews and in person at 12 and 18 months), and by monitoring laboratory parameters at baseline and at 12 months.
Groups:
- Arm A (Aspirin): Participants receive aspirin orally (PO) once daily (QD) for 12 months
Arm/Group | Arm A (Aspirin) | Arm B (Placebo)
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 3/8 | 2/8
Other Adverse Events (participants affected / at risk) | 7/8 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Aspirin) (N=8) | Arm B (Placebo) (N=8)
Subdural Hematoma (Vascular disorders) | 0 | 1
Drainage of Subdural Hematoma (Surgical and medical procedures) | 0 | 1
Parotidectomy (Surgical and medical procedures) | 1 | 0
Small Bowel Obstruction (Gastrointestinal disorders) | 1 | 0
Severe Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Hiatus Hernia Repair (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Aspirin) (N=8) | Arm B (Placebo) (N=8)
Abdominal pain/Abdominal pain with Bloating (Gastrointestinal disorders) | 2 | 0
Acid Reflux (Gastrointestinal disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Blood in Stool (Gastrointestinal disorders) | 0 | 1
Bruising left arm (Skin and subcutaneous tissue disorders) | 0 | 1
Cataract Removed (Eye disorders) | 0 | 1
Chills (General disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1
Cough/Cough due to Cold Symptoms (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Edema-Limbs (General disorders) | 1 | 1
Eye Pain-Herpes Virus Right Eye (Eye disorders) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Fatigue (General disorders) | 0 | 1
Fusion of Right Great Toe Joint (Surgical and medical procedures) | 0 | 1
Ganglion Cyst Left Finger (Musculoskeletal and connective tissue disorders) | 1 | 0
Gout (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 3 | 0
Gastrointestinal Disorders-Other, specify:Mouth Sores (Gastrointestinal disorders) | 1 | 0
Flu like symptoms(Sick/Cough due to cold symptoms/Nasal and chest congestion) (General disorders) | 2 | 1
Nausea/Nausea and Vomiting (Gastrointestinal disorders) | 3 | 0
PSA out of range (Investigations) | 1 | 0
Pain (General disorders) | 0 | 1
Left rotator cuff tear due to fall (Injury, poisoning and procedural complications) | 1 | 0
Surgical and Medical Procedures-Other, specify-Radiation Therapy (Surgical and medical procedures) | 1 | 0
Gastrointestinal Disorders-Other, specify: dental crown recemented (Gastrointestinal disorders) | 1 | 0
Runny Nose (General disorders) | 1 | 0
Sinusitis (Infections and infestations) | 0 | 1
Sinus Surgery for Streptococcus and Staphylococcus Aureus Bacteria Infection (Infections and infestations) | 0 | 1
Small cut/cut on finger taking a long time to heal (General disorders) | 0 | 1
Rotator Cuff Repair (Surgical and medical procedures) | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Diabetes (Metabolism and nutrition disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1
Hematoma (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-03): https://cdn.clinicaltrials.gov/large-docs/85/NCT02521285/Prot_SAP_000.pdf